CLINICAL TRIAL: NCT05530213
Title: Interlaboratory Reliability of 3D Gait Analysis Performed on an Instrumented Treadmill.
Brief Title: Interlaboratory Reliability of 3D Gait Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: Hasselt University (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: ONZ-2022-0248
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Gait Analysis; Reproducibility
Keywords: Norm database; Reliability; 3D gait analysis
MeSH Terms: interventions — Weights and Measures; Body Height

STUDY DESIGN:
Intervention Model Description: A single group of participants will be tested in 3 locations. Their results across the three locations will be compared
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be carried out by investigators who are blind to the location of where the data was collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy adults UZ Gent (Experimental): A group of 30 healthy adults aged 18-65years old will carry out a 3D gait analysis at UZ Gent within a week of the 3D gait analysis at UHasselt and/or UMaastricht.
  Interventions: Device: 3D gait analysis on the GRAIL; Other: Weight and height
- Healthy adults UHasselt (Experimental): The same group of 30 healthy adults aged 18-65years old will carry out a 3D gait analysis at UHasset within a week of the 3D gait analysis at UZGent and/or UMaastricht.
  Interventions: Device: 3D gait analysis on the GRAIL; Other: Weight and height
- Healthy adults UMaastricht (Experimental): The same group of 30 healthy adults aged 18-65years old will carry out a 3D gait analysis at UHasset within a week of the 3D gait analysis at UZGent and/or UZGent.
  Interventions: Device: 3D gait analysis on the GRAIL; Other: Weight and height

INTERVENTIONS:
Device: 3D gait analysis on the GRAIL — 3D gait anlysis performed on an instrumented treadmill (GRAIL, Motek Medical)
Other: Weight and height — The subject's body weight and height will be assessed

SUMMARY:
The purpose of this study is to determine the interlaboratory reliability of 3D gait analysis performed on healthy subjects on an instrumented treadmill in three different laboratories. This will allow us to evaluate whether the pooling of control data is feasible in future studies. This will support our ambitions to enter into future collaborations to conduct studies with larger samples. Moreover, this way we will know if we can share patient data in the future so that patients can be specifically referred to a lab with expertise on a particular evaluation, e.g. the lab in Maastricht has expertise on perturbations, UZ Gent has expertise on full-body measurements and UHasselt has expertise on balance.

During this study approximately 30 healthy subjects will be recruited (10 from each center) from the staff and students at each center. These subjects are own staff and students of the 3 centers. Each subject will undergo a 3D gait analysis at each center (at UZGent, UHasselt and UMaastricht). Therefore, each subject will be evaluated 3 times. The time between each evaluations will be a maximum of one week.

The evaluations will be performed as per standard procedure in each lab. However, a standardized model (HBM2 lower limb), an agreed walking velocity (0.9 m/s, 1.0 m/s, 1.1 m/s) and an agreed duration per recording (3 min) will be used. The same software will be used to process the collected data. 3D kinematics and kinetic time-series data of the lower limbs will be extracted as outcome data. Absolute reliability indices will be calculated in the following way: First, the standard deviation (SD) of time-series data across different gait cycles will be calculated per participant per center. The SD values across different centers per participant will then be averaged. Finally, the SD values across different participants will form the inter-laboratory reliability indices. In addition, we will use statistical parametric mapping (Anova repeated measures) to compare the full time-series data of each outcome parameter.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects aged 18-65 years old

Exclusion Criteria:

Individuals cannot participate if:

* They suffer from a neurological disorder.
* They experience balance problems.
* They have had surgical procedures on the legs in the past.
* They are taking medication that may affect gait and balance. They experience leg or back pain at the time of test taking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
3D lower limb kinematics (angles °) | Single point of assessment in one day
  Marker trajectory data is collected during the 3D gait analysis and lower limb kinematics are calculated in post-processing. Pelvis, hip, knee and ankle angles will be assessed during walking at 3 different gait velocities
3D lower limb kinetics (Nm/kg) | Single point of assessment in one day
  Force plate data is collected during the 3D gait analysis and hip, knee and ankle kinetics are calculated while walking at 3 different gait velocities.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Bar-On, PhD, Principal Investigator — UGent
Locations (2):
- University Hasselt, Hasselt, Belgium
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the ethics agreements, an IPD data sharing plan document is available at each institute.
Supporting Information: Study Protocol, SAP, Analytic Code